CLINICAL TRIAL: NCT00520637
Title: A Phase I, Multicenter, Open-Label, Dose-Escalation Study Evaluating the Safety and Tolerability of Intravenous EZN-2208 (PEG-SN38) Administered Every 3 Weeks in Patients With Advanced Solid Tumors or Lymphoma (EZN-2208-01)
Brief Title: A Phase I, Study to Evaluate the Safety and Tolerability of Intravenous EZN-2208 in Patients With Advanced Solid Tumors or Lymphoma (EZN-2208-01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: EZN-2208-01
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Advanced Solid Tumors; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — EZN-2208

INTERVENTIONS:
Drug: EZN-2208

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of EZN-2208 that can be given to patients with advanced cancer or lymphoma. The safety of the study drug and its effect on the disease will also be studied.

Enzon will also perform pharmacokinetic (PK) testing of EZN-2208. PK testing measures the amount of a drug in the body at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced and/or metastatic solid tumor or lymphoma that is refractory to standard therapy
* Measurable or evaluable disease
* Score of 0 to 2 on the ECOG performance scale

Exclusion Criteria:

* Concurrent serious medical illness
* Known, clinically suspected, or history of central nervous system (CNS) tumor involvement
* Active diarrhea
* Known history of coagulation disorder
* Patients requiring cytochrome P450 3A4 (CYP3A4) enzyme inducing medications
* Requirement for ketoconazole or other strong inhibitor of CYP3A4 enzymes
* Prior chemotherapy, immunotherapy, investigational agent, or other therapy used to treat the cancer within 4 weeks (6 weeks for prior treatment with mitomycin C or nitrosoureas) prior to the scheduled administration of EZN-2208

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2007-05

PRIMARY OUTCOMES:
Determine the MTD of i.v. EZN-2208 administered q3wk and recommended Phase 2 dose of i.v. EZN-2208

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of EZN-2208, assess the pharmacokinetic PK profile of EZN-2208, SN38, and SN38G as well as detect preliminary evidence of tumor response activity of EZN-2208

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, MD, Principal Investigator — M.D. Anderson Cancer Center; Mary Frances Mulcahy, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (2):
- United States (2):
  - Northwestern University, Feinberg School of Medicine, Division of Hematology/Oncology, Chicago, Illinois
  - MD Anderson Cancer Center, Houston, Texas